CLINICAL TRIAL: NCT04699513
Title: The Effect of Preemptive Airway Pressure Release Ventilation on Patients With High Risk for Acute Respiratory Distress Syndrome: a Randomized Controlled Trial
Brief Title: The Effect of Preemptive APRV on Patients With High Risk for ARDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Collaborators: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, mehtap pehlivanlar küçük, Consultant Intensivist, Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2016/175
Record Dates: First submitted 2021-01-04; First posted 2021-01-07 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Acute Respiratory Distress Syndrome; Intensive Care Unit
Keywords: APRV; Intensive Care Unit
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Intervention Model Description: a randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- P-SIMV+PS group (Experimental): The reason behind using P-SIMV+PS as a conventional mode was that it is a pressure controlled mode like APRV.
  Interventions: Device: Mechanical Ventilation Mode (airway pressure release ventilation )
- APRV group (Experimental): Airway pressure release ventilation (APRV) is a mode of mechanical ventilation that alternates between two levels of continuous positive airway pressure (CPAP) support and allows spontaneous respiratory effort at either CPAP level. It is considered as an alternative, life-saving modality in patients with acute respiratory distress syndrome (ARDS) that struggle for oxygenation.
  Interventions: Device: Mechanical Ventilation Mode (airway pressure release ventilation )

INTERVENTIONS:
Device: Mechanical Ventilation Mode (airway pressure release ventilation ) — Airway pressure release ventilation (APRV) is a mode of mechanical ventilation that alternates between two levels of continuous positive airway pressure (CPAP) support and allows spontaneous respiratory effort at either CPAP level. It is considered as an alternative, life-saving modality in patients with acute respiratory distress syndrome (ARDS) that struggle for oxygenation.

SUMMARY:
Airway pressure release ventilation (APRV) is a mode of mechanical ventilation that alternates between two levels of continuous positive airway pressure (CPAP) support and allows spontaneous respiratory effort at either CPAP level. It is considered as an alternative, life-saving modality in patients with acute respiratory distress syndrome (ARDS) that struggle for oxygenation. Compared to the classical ventilation, APRV has been shown to provide lower peak pressure, better oxygenation, less circulatory loss, and better gas exchange without deteriorating the hemodynamic condition of the ARDS patient. This mode is believed to help to achieve the target of opening consolidated lung areas (recruitment) and to prevent repeated opening-closing of alveoli (decruitment). However, there is still insufficient and limited proof to support this hypothesis.

Recently, it has been proposed that early use of protective mechanical ventilation with APRV could be used preemptively to prevent development of ARDS in high risk patients. In that study, APRV prevented clinical and histological lung injury by protecting alveolar epithelial integrity, preserving surfactant and alveolar stability, and reducing pulmonary edema.

The primary purpose of the present study was to investigate whether early use of APRV as a lung-protecting strategy was superior to the conventional methods in a patient population with high risk of acute respiratory distress syndrome (ARDS).

DETAILED DESCRIPTION:
This study was planned as a single-centered, prospective, and randomised-controlled study in a general intensive care unit with 18 bed capacity. The majority of the general patient population is made up of trauma and post-operative patients. The local ethics committee reviewed and approved the study protocol (protocol number: 2016/175) prior to the start of the investigation. Enrollment for the study was performed between May 2016-October 2018. Written informed consent was obtained from each patient's relatives.

Study design and sample:

The study included patients who required invasive mechanical ventilation but was not initially diagnosed with ARDS 9, had a LIPS (Lung Injury Prediction Score) of > 7 10, and have been staying in the ICU for more than 24 hours. Patient demographic properties, sedation requirements, inotrope/vasopressor levels, ARDS development status during follow-up, mechanical ventilation times, length of ICU stay, arterial blood gas results, mean airway pressure (Pmean), peak airway pressure (Ppeak) and tidal volume (Vt) in addition to the mode-specific mechanical ventilation parameters were recorded. Exclusion criteria were pregnancy, intracranial hypertension (suspected or confirmed by measurement with external ventricular drainage catheter), severe chronic obstructive pulmonary disease or type II respiratory failure, confirmed bronchopleural fistula, documented barotrauma, history of pneumonectomy, and age below 18 or above 85 years. Consecutive eligible patients were enrolled block randomization with a 1:1 allocation, randomly assigned to APRV or P-SIMV+PS groups using opaque, sealed envelopes.

Ventilator Settings:

All mechanical ventilation settings were made by intensivists, or trained residents on the night shifts. Prior to randomization, all patients were treated with VC-SIMV mode. Patients admitted during the day were ventilated in VC-SIMV mode until the main investigators evaluated the patient (1-2 hours), and patient admitted in the evening-night shift were ventilated in VC-SIMV mode until the main investigators took over the shift in the morning (maximum 16 hours). Assignment to groups was performed after calculation of LIPS score. Microprocessor-controlled mechanical ventilators (Galileo GOLD; Hamilton Medical AG, Bonaduz, Switzerland) and heated humidifiers were used as a standard in all patients. In both groups, mechanical ventilation targets were determined as maintaining plateau airway pressure (Pplateu) < 30 cmH2O and PaO2 between 60-100 mmHg or SO2>88%. In both groups, arterial blood gas measurement was performed at least twice a day. Oxygenation and respiratory mechanics were evaluated by comparing P-SIMV+PS and APRV groups at baseline and on days 1, 2, 3, and 7. Patients were followed until transfer to CPAP/T-tube and extubation, or a maximum of 28 days. During this period, follow-up was terminated once at extubation, exitus, discharge from ICU or ARDS occurred.

P-SIMV+PS group:

The reason behind using P-SIMV+PS as a conventional mode was that it is a pressure controlled mode like APRV. Pressure level was adjusted in order to get a Vt of 6-8 ml.kg-1.PBW-1 (predicted body weight). Optimal PEEP between 5-10 cmH2O was applied to all patients by titrating according to O2 requirement. Respiratory rate was adjusted as 12-15 breaths.min-1, and inspiratory time was initially adjusted to approximately 1.5 seconds. The I:E ratio was adjusted by either changing inspiratory time, respiratory rate, or both. Inspiratory triggering sensitivity was adjusted as 2 L.min-1, and was tittered by reaching the minimum level in the absence of automatic triggering.

APRV group:

Standard initial settings were Thigh / Tlow: 4/0.8 secods, Phigh: taking Pplateau value (if patient is paralyzed) or Pmean in the previous conventional method as reference, Pplateau < 30 cmH20 and target Vt 6-8 ml.kg-1.PBW-1. Plow was always set to 0 cmH2O. T-low was adjusted according to PCO2 value in blood gas measurement, by evaluating expiratory flow curve (gas flow wave form), and to get a release duration of 10-14.cycle-1. Tlow range was adjusted as 0.4-1.2 seconds. When needed, Thigh was gradually increased to 12-15 seconds by increments of 1-2 seconds. In case of hypoxemia, the problem was generally solved by increasing Phigh and FiO2, and as an additional strategy, Thigh was increased. In case of hypercapnia, sedation was lowered to allow spontaneous breaths. In order to increase the number of releases and thus, increase the minute-ventilation, Thigh was shortened and Phigh was increased 12,13.

Weaning Process:

Weaning was performed according to the European Respiratory Society Weaning Task Force recommendations in both groups 14. In APRV group, Phigh was reduced by 2-3 cmH2O and Thigh increased by 0.5-2.0 sec during weaning as the patient tolerated it. Tlow was kept constant at the same time. Before transfer to CPAP, Phigh was kept at approximately 14-16 cm H2O or lower, and Thigh was increased up to level of 10-12 sec. In P-SIMV+PS group, respiratory rate was reduced by 2 breaths.min-1, and PS level was reduced by decrements of 2-4 cmH2O. In both groups, spontaneous breathing trial was attempted for 30-60 minutes with T-tube when CPAP was 5-10 cmH2O, and patients were extubated afterwards. For patients with tolerance, the same trial was repeated the next day. Total MV time was defined as the time passed from intubation to the last successful extubation. Patients who required tracheotomy during follow-up were recorded.

Medical and Supportive Treatments:

Preferred medications for those patients requiring sedation was midazolam infused at loading dose: 0.5 to 5 mg every 1 to 5 minutes (if needed), followed by 1 to 8 mg.hour-1 or 0.01 to 0.1 mg.kg-1.hour-1 continuous infusion; titrate infusion rate to clinical effect; for analgesia, fentanyl infused at 1-2 mcg.kg-1.hr-1 i.v. The sedation goal was a Richmond Agitation Sedation Scale score of - 2 to 0 15. According to our clinic's sedation policy, Richmond Agitation Sedation Scale was assessed hourly by the nursing staff, and medication doses were titrated by the respiratory therapists according to target spontaneous respiration level. Evaluation of whether patients received sedation and the number of days which they received sedation were recorded. Sedation doses were not evaluated. None of the patients received neuromuscular blocker. Fluid management, antibiotic strategy, glucose control and enteral nutrition were also standardized between the two groups according to the ICU protocols.

Statistical Analysis On the primary outcome of developing ARDS in the light of P/F ratio 8[Clinically defined ALI/ARDS developed in the CMV group (mean [SE] PaO2/FIO2 [P/F] ratio, 242.96 [S.E. 24.82]), and this was prevented with APRV (P/F ratio, 478.00 [S.E.41.38]; P < .05 vs CMV)], power analysis using the Gpower computer program11 indicated that a total sample of 58 people would be needed to detect large effects (d: 0.888) with 90% power using a t test between means with 2-tailed alpha at .05.

All data were analyzed using IBM SPSS V23 (Chicago, USA). The Shapiro Wilk test was used to determine whether the data were normally distributed. Comparisons of data that were not normally distributed were made with the Kruskal Wallis test and the Mann Whitney U test. Categorical data were analyzed with the Pearson chi-square test. The groups were compared with regard to laboratory parameters measured on days 1, 2, 3, and 7. Non-normally distributed data were presented as median (min-max), while normally distributed data were presented as mean ± standard deviation. Categorical data were expressed as frequency and percentage. Values of p < .05 were considered significant.

Study Endpoint The primary endpoint of the study was to determine whether APRV mode was protective against ARDS compared to the conventional mode in patients with high risk of ARDS as determined by LIPS score. The secondary endpoint was to determine whether this mode provided any improvement in oxygenation, airway pressures, sedation and inotrope requirements, mechanical ventilation time and length of ICU/hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* The study included patients who required invasive mechanical ventilation but was not initially diagnosed with ARDS 9, had a LIPS (Lung Injury Prediction Score) of > 7, and have been staying in the ICU for more than 24 hours.

Exclusion Criteria:

* pregnancy
* intracranial hypertension (suspected or confirmed by measurement with external ventricular drainage catheter)
* severe chronic obstructive pulmonary disease or type II respiratory failure
* confirmed bronchopleural fistula
* documented barotrauma
* history of pneumonectomy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
ARDS | 2 year
  Early use of APRV as a lung-protecting strategy was superior to the conventional methods in a patient population with high risk of acute respiratory distress syndrome (ARDS)
P/F ratio | 2 year
  Affect of early using of APRV on P/F ratio, as a lung-protecting strategy was superior to the conventional methods in a patient population with high risk of acute respiratory distress syndrome (ARDS)

SECONDARY OUTCOMES:
Mortality | 2 year
  The secondary endpoint was to determine whether this mode provided any improvement in mortality of ICU.
Oxygenation | 2 year
  The secondary endpoint was to determine whether this mode provided any improvement in oxygenation by assessing partial pressure of oxygen in artery blood gas.
Airway pressures | 2 year
  The secondary endpoint was to determine whether this mode provided any improvement in airway pressures (mean airway pressure (Pmean), peak airway pressure (Ppeak)).
Sedation requirements | 2 year
  The secondary endpoint was to determine whether this mode provided any improvement in sedation requirements (% of present in the population).
inotrope requirements | 2 year
  The secondary endpoint was to determine whether this mode provided any improvement in inotrope requirements (% of present in the population).
Mechanical ventilation duration in the ICU | 2 year
  The secondary endpoint was to determine whether this mode provided any improvement in mechanical ventilation duration (day) in the ICU .
Mechanical ventilation time and length of ICU/hospital stay. | 2 year
  The secondary endpoint was to determine whether this mode provided any improvement in length of ICU/hospital stay (day).

CONTACTS AND LOCATIONS:
Overall Officials: Mehtap Pehlivanlar Küçük, MD, Study Chair — Karadeniz Technical University, Faculty of Medicine

IPD SHARING:
Plan to Share IPD: No